CLINICAL TRIAL: NCT04141761
Title: Probiotic-induced Normalization of Innate Inflammation in Youth Newly Diagnosed With Type 1 Diabetes
Brief Title: Probiotics in Newly Diagnosed T1D
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Susanne Cabrera, Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1343363
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes; Type1diabetes; Type 1 Diabetes Mellitus
Keywords: Newly diagnosed; Recent onset; Visbiome; Probiotic
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single-blind, placebo-controlled, 2:1 randomly assigned
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Dietary Supplement: Visbiome
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Visbiome — This group will receive Visbiome probiotic in powder form.
  Arms: Treatment Group
Other: Placebo — This group will receive a placebo in powder form.
  Arms: Placebo Group

SUMMARY:
The investigators aim to further the understanding of environmental factors that underlie the development of Type 1 diabetes (T1D) and the post-onset disease trajectory. Dysbiosis, defined as alterations in intestinal microbiota composition and function, has been hypothesized to increase the risk of developing T1D in those with genetic susceptibility. Dysbiosis may result from modern dietary habits, such as broad consumption of the highly processed Western Diet, or by widespread use of antibiotics. Here, the investigators propose to examine the impact of dysbiosis on the endogenous innate inflammatory state that potentiates T1D progression. The investigators hypothesize that probiotic-induced alterations in the intestinal microbiota may favorably alter the post-onset disease state.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria:

  1. Males and females 5-17 years of age with a clinical diagnosis of T1D within the past 90 days
  2. Positive for ≥ 1 diabetes-related autoantibodies (IAA, GAD, IA-2, or ZnT8)
  3. Stimulated C-peptide area under the curve (AUC) of ≥ 0.2 nmol/L during a mixed meal tolerance test
  4. Treatment naïve of any immunomodulatory agent

Exclusion Criteria:

* Patients must NOT meet any of the following criteria:

  1. Probiotic use within 1 month of screening visit
  2. Presence of severe, active disease that requires the use of chronic medication, with the exception of well-controlled autoimmune thyroiditis/hypothyroidism
  3. Diabetes other than T1D
  4. Female participants of child-bearing age with reproductive potential must not be knowingly pregnant
  5. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Multistrain Probiotic on Immune System Inflammation as measured by plasma transcription analysis | 3 years (duration of study)
  Investigators will examine the effect of multistrain probiotic supplementation on the endogenous innate inflammatory state in youth newly diagnosed with T1D, as measured by plasma-induced transcription analysis. The investigators hypothesize that the participants receiving the probiotic will have less inflammation (as measured by transcriptional analysis) than the participants in the placebo group.

SECONDARY OUTCOMES:
C-peptide decline | 3 years (duration of study)
  Investigators will examine the effect of multistrain probiotic supplementation on the post-onset rate of C-peptide decline (a measure of beta cell health)
Effect of Multistrain Probiotic on broader Immune System Effects as measured by plasma-induced transcriptional analyses | 3 years (duration of study)
  Investigators will examine the effect of multistrain probiotic supplementation on changes to the plasma-induced transcriptional assay to assess for probiotic-specific immune effects. Plasma-induced transcriptional analyses will be compared before and after treatment with probiotic/placebo. The investigators hypothesize that the participants receiving the probiotic will see reduced inflammation (as measured by transcriptional analysis) while those that received the placebo will see no change or increased inflammation.
Cytokine Levels (a measure of inflammation) as measured by plasma analysis | 3 years (duration of study)
  Cytokine levels before and after treatment will be measured by plasma analysis. It is hypothesized that the levels of cytokines in the blood will be lower after treatment for the participants receiving the probiotic but not for those receiving the placebo.
Changes to intestinal bacteria as measured by stool analysis | 3 years (duration of study)
  Investigators will examine the effect of multistrain probiotic supplementation the composition of the intestinal microbiota
System-wide Effects as measured by systemic microbial antigen (a marker of intestinal permeability) as measured by plasma analysis | 3 years (duration of study)
  Gut leakiness will be measured by examining the levels of microbial antigens in the plasma before and after treatment and correlating these antigen levels with the changes in the composition of the gut bacteria. It is hypothesized that changes in antigen levels and gut bacteria will only be seen in the participants receiving the probiotic. It is further hypothesized that those with the greatest reduction in antigens will have the most significant changes in gut bacteria composition.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No